

Statistical Analysis Plan

Phase I clinical study, to evaluate the safety and tolerability of PRO-165 ophthalmic gel versus Artelac® Nightime Gel, on the ocular surface of ophthalmologically and clinically healthy subjects.



Date of creation: July 2017.

Phase I clinical study, to evaluate the safety and tolerability of PRO-165 ophthalmic gel versus Artelac® Nightime Gel, on the ocular surface of ophthalmologically and clinically healthy subjects.

Protocol Code: SOPH165-0217/I.

Protocol Version: 2.0

### Content

| 1.0 | Abbreviations | 3 | |
|-----|-----------------------------|----|---|
| 2.0 | Objectives of the Study | 3 | |
| 3.0 | Study Design SOPH165-0217/I | 4 | |
| 4.0 | Sample Size | 5 | |
| 5.0 | Sample Size Calculation | 6 | |
| 7.0 | Methods of Analysis | 11 | |
| 8.0 | Changes | 15 | |
| 9.0 | References | 13 | 5 |
| 100 | Annexes | 16 | |

### **Abbreviations**

BHc Complete hematic biometry

CRF Electronic Case Report Form

VA Visual Ability

AE Adverse events

HR Heart rate

FCI Informed Consent Form

FR Respiratory rate

HC Conjunctival hyperemia

ICO Eye Comfort Index

ITT Population by intent to treat

SC Safety call

MC Concomitant medication

PFH Liver function tests

RP Research Product

IOP Intraocular pressure

PP Population by protocol

PRO-165 Chondroitin sulfate 0.18%/Sodium hyaluronate 0.2%

BC Blood chemistry

SBP Systemic blood pressure

TBUT Tear break-up time

BV Initial visit FV Final visit

# Objective of the Study

To evaluate the safety and tolerability of the PRO-165 formulation on the ocular surface of ophthalmologically and clinically healthy subjects.

# Study Hypothesis

H0: PRO-165 Ophthalmic Gel has a similar safety and tolerability profile to Artelac® Nightime Gel in ophthalmologically and clinically healthy subjects.

H1: PRO-165 Ophthalmic Gel has a different safety and tolerability profile than Artelac® Nightime Gel in ophthalmologically and clinically healthy subjects.

# Study Design SOPH165-0217/I

Phase I, controlled, parallel-group, double-blind, randomized, exploratory clinical trial.

### Duration of treatment

Treatment: 10 days.

Study period: 4 months.

Table 1. Study timeline

| Procedures | Scrutiny | Basal<br>Visit | Visit 1 | Final Visit | Call<br>Security |
|---|---|---|---|---|---|
| Procedures | Day 0 - X <sup>to</sup> | Day 0 | Day 5 ± | Day 11 to<br>+ 1 | Day 13 ± 1 |
| CI Signature | Х | | | | |
| Medical history | X | | | | |
| Ophthalmological medical history | Х | | | | |
| Laboratory sample collection | Х | | | Х | |
| Review of Laboratory Tests | | Х | | | Х |
| Pregnancy Test | Х | | | X | |
| Eligibility Criteria | Х | Xb | | | |
| Allocation | | Х | | | |

Chondroitin Sulfate 0.18%/Sodium Hyaluronate 0.2%

| Delivery of intervention | | Xc | | | |
|----------------------------------------------------|---|-----|---|---|---|
| Return of intervention | | | | Х | |
| Adherence assessment | | | Х | Х | |
| Adverse events | | | Х | Х | Х |
| Intraocular pressure | X | 1 x | Х | Х | |
| Visual Ability | X | 1 x | Х | Х | |
| TRL | X | 1 x | Х | Х | |
| Ocular surface stains | X | 1 x | Х | Х | |
| Vitals | X | 1 x | Х | Х | |
| Eye Comfort Index | | Х | | Х | |
| Subject Diary Delivery | | Х | Х | | |
| Return / Evaluation of the subject's Journal | | | Х | Х | |
| Return and Evaluation of the Quality Questionnaire | | | | Х | |
| Subject continuity assessment | | | Х | | |

<sup>&</sup>lt;sup>a</sup> The counting visit may be up to 10 days prior to the baseline, if it exceeds these the subject will not be able to enter.

# Sample Size

An estimated 32 evaluable subjects are divided, divided into two groups [16 subjects (16 eyes) exposed per group].

<sup>&</sup>lt;sup>b</sup> These criteria shall be supplemented by the results of laboratory examinations and those collected during the screening visit.

<sup>&</sup>lt;sup>c</sup> An indication will be given to start the application the next day.

<sup>&</sup>lt;sup>1</sup>They can be taken from the scrutiny visit, as long as no more than 10 days have elapsed, it is the prerogative of the PI to measure them again at the baseline visit.



Figure 1. Suggested work scheme.

### Sample Size Calculation

There are no references to sample size calculation in phase I studies, and the formulation of Humylub Ofteno® has not reported adverse events in its periodic safety reports. For this reason, it was considered pertinent to base it on the calculations of previous phase I studies, carried out by Laboratorios Sophia, S.A. de C.V., with formulations of ocular lubricants in the same pharmaceutical presentation.

The calculation was in accordance with the presentation of adverse events reported by Christ T (1994), in a randomized, single-blind, parallel-group controlled clinical trial where the efficacy and tolerance of a 5% dexpanthenol ophthalmic gel versus a 5% panthenol ointment in 48 subjects with corneal erosion was evaluated. keratoconjunctivitis from UV radiation or similar conditions. The intervention consisted of the application of 1 cm of the gel and ointment for 4 and 3 days, respectively. [1][2]

The percentage of good tolerance that was presented with the gel was 25%, so it is expected that no more than 10% of the subjects report a bad tolerance with the formulation proposed in this protocol.

The sample size was calculated using the formula for proportions.[3]

$$n = p(1-p) \left(\frac{z_{1-\alpha} + z_{1-\beta}}{p - p_0 - \delta}\right)^2$$

With a statistical confidence of 95% that corresponds to type I error, equal to 1.96, with a power of 90%, corresponding to type II error, equal to 0.84.

According to the previous calculation, the result is 26 subjects, which was increased by 20% due to the probable losses. The total sample size required is 32 subjects. So each group will be made up of 16 subjects, who will provide an eye for the analysis.

# Analysis Plan [4]

### **Outcome Variables**

Safety primary outcome variables:

Incidence of Adverse Events.

Primary outcome variables of tolerability:

ICO score.

### Secondary Outcome Variables:

- Tear film rupture time (LRT).
- Vital signs: HR, RF and SAP.
- Posterior segment.
- Quality questionnaire.
- Intraocular pressure.
- Visual capacity.
- Laboratory Tests: BHc, QS, PFH.
- Ocular surface stains.

# Table 2. Operational Definition of the Variables

| Variable | Conceptual<br>Definition | Operational<br>Definition | Measurement<br>Type | Normal value | Statistical<br>test |
|---|---|---|---|---|---|
| Adverse<br>events (AEs). | Any undesirable medical event that may occur in an investigational subject during the clinical research stage of a drug or vaccine but does not necessarily have a causal relationship with it.4 | Adverse events<br>manifested during<br>the conduct of the<br>study will be<br>collected using the<br>CRF. | - Continuous quantitative Categorical qualitative. | - Frequency: Subjects with AEs/Total number of exposed subjects. - Intensity: 0= Mild 1= Moderate 2= Severe - Causality: 0= Improbably related. 1= Probable or possibly related. 2= Related | - Pearson's square chi or Fisher's exact U for Mann-Whitney. |
| Changes in<br>Intraocular<br>Pressure<br>(IOP). | Tonometry is the objective measurement of IOP, based primarily on the force required to flatten the cornea or the degree of corneal indentation produced by a fixed force. | Goldmann<br>tonometry. 3 samples<br>will be taken, which<br>will be recorded in<br>the clinical file and<br>the average will be<br>recorded in the CRF. | - Continuous<br>quantitative. | - 11-21 mmHg. | - U for<br>Mann-<br>Whitney.<br>- Wilcoxon<br>Ranges. |
| Eye Comfort<br>Index (ICO)<br>score. | The ICO is a questionnaire designed to measure irritation of the ocular surface, it assesses symptoms | The evaluator will apply the questionnaire to the subject and allow the subject to answer it calmly without any pressure and/or | Discrete<br>quantitative. | Score: 0= None, 100 = High discomfort. | - U for<br>Mann-<br>Whitney.<br>- Wilcoxon<br>Ranges. |

| | focused on the comfort associated with ocular surface alterations. Elevated values indicate more Severe. | coercion. See ICO<br>Annex. | | | |
|---|---|---|---|---|---|
| Changes in visual capacity (CV) | Visual acuity (VA) is a test of visual function. Spatial VA is the ability to distinguish separate elements of an object and identify them as a whole. It is quantified as the minimum angle of separation (located at the nodal point of the eye) between two objects that allows them to be perceived as separate objects. | Snellen's Primer | Discrete<br>quantitative. | Fraction, normal<br>value = 20/20 | - U for<br>Mann-<br>Whitney.<br>- Wilcoxon<br>Ranges. |
| Changes in<br>tear film<br>rupture time<br>(LRT) with<br>fluorescein. | The stability of the tear film is usually evaluated in the clinic by the TRL. It consists of instilling fluorescein on the ocular surface to allow the visualization of the tear film | It will be measured at the end of a blink and will be asked not to blink immediately until the tear film on the cornea is broken. | Continuous<br>quantitative. | > 10 seconds. | - U for<br>Mann-<br>Whitney.<br>- Wilcoxon<br>Ranges. |

| | and measure<br>the time it<br>takes to break<br>since the last<br>blink. | | | | |
|---|---|---|---|---|---|
| Changes in corneal and conjunctival staining with lysmine green. | Detection of epithelial defects in the conjunctiva and cornea. | Direct observation<br>with slit lamp, Oxford<br>scale graduation. See<br>annex Oxford scale. | Ordinal<br>Qualitative | Degrees: The staining is presented by a series of panels (A-E). Stain points range from 0-5 for each panel and 0-15 for the total exposed area of the conjunctiva and cornea. | <ul> <li>Pearson's square chi or Fisher's exact.</li> <li>McNemar test (if applicable).</li> </ul> |
| Corneal and conjunctival staining changes with fluorescein. | Detection of epithelial defects in the conjunctiva and cornea. | Direct observation<br>with slit lamp and<br>cobalt blue filter,<br>Oxford scale<br>graduation. See<br>annex Oxford scale. | Ordinal<br>Qualitative | Degrees: The staining is presented by a series of panels (A-E). Stain points range from 0-5 for each panel and 0-15 for the total exposed area of the conjunctiva and cornea. | <ul> <li>Pearson's square chi or Fisher's exact.</li> <li>McNemar test (if applicable).</li> </ul> |
| Incidence of<br>alterations in<br>laboratory<br>test results. | The normal parameters to be considered will be the ranges established by the laboratory, with a lower and upper margin of 20% in a clinically healthy subject, according to the Pl's criteria. | Laboratory analysis. | Continuous<br>quantitative. | See annex Scales<br>to be used for<br>vital signs and<br>laboratory<br>analysis. | <ul> <li>U for<br/>Mann-<br/>Whitney.</li> <li>Wilcoxon<br/>Ranges.</li> </ul> |

| | | | | _ | |
|---|---|---|---|---|---|
| Incidence of<br>alterations in<br>HR. | The normal parameters to be considered will be the ranges established by the laboratory, with a lower and upper margin of 20% in a clinically healthy subject, according to the PI's criteria. | Auscultation with a stethoscope. | Continuous<br>quantitative. | 60-100 lpm. | - U for Mann-<br>Whitney.<br>- Wilcoxon<br>Ranges. |
| Incidence of<br>alterations in<br>RF. | The normal parameters to be considered will be the ranges established by the laboratory, with a lower and upper margin of 20% in a clinically healthy subject, according to the PI's criteria. | Auscultation with a stethoscope. | Continuous<br>quantitative. | 12-24 rpm. | - U for Mann-<br>Whitney.<br>- Wilcoxon<br>Ranges. |
| Incidence of<br>abnormalities<br>in SBP. | The normal parameters to be considered will be the ranges established by the laboratory, with a lower and upper margin of 20% in a clinically healthy subject, according to the Pl's criteria. | Measurement with sphygmomanometer. | Continuous<br>quantitative. | < 120 / 80<br>mmHg | - U for Mann-<br>Whitney.<br>- Wilcoxon<br>Ranges. |

# Methods of Analysis [4]

The statistical analysis will be carried out by personnel of Laboratorios Sophia, S.A. de C.V. The statistical program SPSS version 19.0 (IBM Corporation, Armonk, NY, USA) will be used. Designated personnel will be blinded to intervention groups. Coding will be performed using consecutive numbers for each intervention group.

The data will be collected and sorted in an Excel spreadsheet (Microsoft® Office). The data will then be exported to the SPSS program platform. The variables will be categorized according to their nature (see Table 2).

Study participants will be identified by a number and their initials.

The initials of the study subject will be obtained starting with the first letter of the name, followed by the first letter of the first surname and the first letter of the second surname, obtaining a maximum of three letters, in case the person has two names or compound surname, the first letter will always be used.

### Example:

#### To. Arieh Daniel Carrizalez Market

B. Juan De la Torre Orozco

to. Initials: AMC

b. Initials: JDO

Once the subject has been selected, they will be assigned a number with which they will be identified throughout the study. This code will be made up of eight numbers in the following order from left to right:

- Three digits of the molecule under study according to the name by the sponsor.
- Two digits corresponding to the research centre number.
- Three digits of the number following their inclusion assigned to the research centre.

The results of the continuous quantitative variables will be presented in measures of central tendency: mean, standard deviation and ranges, see Table 2.

The Kolmogorov-Smirnov and Shapiro Wilk test will be performed to determine the type of distribution of the data (normality) in the results obtained in each study group. [5]

The statistical analysis of the continuous quantitative variables to find significant differences (p) will be as follows:

- <u>Intra-group analysis:</u> will be determined by Wilcoxon's rank test, for quantitative variables. [6]
- <u>Inter-group analysis:</u> Differences between groups will be analyzed using the Mann-Whitney U statistic.

The level of difference to consider significance will be an alpha ( $\alpha$ ) of 0.05 or less. A 95% CI will be considered for the non-inferiority criteria.

The result of the nominal and ordinal qualitative variables will be presented in frequencies, proportions and percentages, see Table 2.

The statistical analysis to identify significant differences in the qualitative variables will be carried out by creating 2x2 contingency tables and will be carried out as follows:

- <u>Intra-group difference</u>: McNemar test. This is applied to 2×2 contingency tables with a dichotomous feature, with pairs of paired subjects, to determine if the marginal frequencies of row and column are equal (marginal homogeneity).
- <u>Difference between groups:</u> Pearson's Chi-square (*X2*) test or Fisher's exact test at expected values less than 5.

The level of difference to consider significance (p) will be an alpha ( $\alpha$ ) of 0.05 or less.

For the reporting of adverse events, all eyes of those participants who were randomly assigned to an intervention group after PI instillation (ITT) will be considered.

The final report of the results will be shown in tables or graphs, as appropriate.

Those subjects who meet a minimum adherence of 60% will be included in the statistical analysis to meet the objective of the study, taken from the subject's diary. However, even if the subject's adherence is greater than 60% per diary, if the adherence calculated by weight is less than 30%, the subject will not be included.

The investigational drug will be considered safe and tolerable when there are no clinical and statistical differences in all primary outcome variables, with respect to its comparator (Artelac® Nightime Gel).

Table 3. Triangulation of concepts

| Variable<br>Type | Variable | <b>A</b> 1 | В1 | B2 | C1 | Dì | E1 | E2 | E3 | E4 | E5 | E6 | E7 | E8 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Backgroun | Background | | | | | | | | | | | | | |
| A1 | Demographic | DT | | | | | | | | | | | | |
| Basal | | | | | | | | | | | | | | |
| B1 | Medical History | DT | | | Т | | | | | | | | | |
| B2 | Comprehensive ophthalmological evaluation | DT | DT | | ТВ | | | | ТВ | | В | В | | Т |
| Safety | | | | | | | | | | | | | | |
| C1 | Incidence of AD | | | ТВ | ТВ | | ТВ | ТВ | ТВ | | ТВ | ТВ | ТВ | ТВ |
| Tolerability | , | | | | | | | | | | | | | |
| D1 | ICO | DB | | | | DB | | | | | | | | |
| Secondary outcome | | | | | | | | | | | | | | |
| E1 | TRL | DB | | | ТВ | | DB | | | | | | | |
| E2 | Vitals | DB | | | ТВ | | | В | | | | | | |

| E3 | Posterior segment | | DB | ТВ | В | | | |
|---|---|---|---|---|---|---|---|---|
| E4 | Quality Questionnaire | | | | Т | В | | |
| E5 | PIO | | DB | ТВ | | В | | |
| E6 | Visual Ability | | DB | ТВ | | В | | |
| E7 | Laboratory tests | DB | | ТВ | | | В | |
| E8 | Ocular surface stains | | ТВ | ТВ | | | | ТВ |
| D, Descri | D, Descriptive Statistics; T, 2x2 contingency table; B, Bivariate Analysis; M, Multivariate Analysis. | | | | | | | |

# Changes

1. First version of the document, no changes apply.

### Author of the document

Ph.D. in Cs. Patricia Muñoz Villegas.

Biostatistics.

Clinical Operations.

Laboratorios Sophia, S.A. de C.V.

Av. Paseo del Norte 5255, Guadalajara Technology Park.

45010, Zapopan, Jalisco, Mexico.

# References

- 1. Christ T. Christ, T. Spektrum Augeheilkd (1994) 8: 224. https://doi.org/10.1007/BF03163747.
- 2. Laboratorios Sophia, SA de CV., National Registry of Clinical Trials (RENEC). [Online] Available:

http://189.254.115.252/Resoluciones/Consultas/ConWedRegEnsayosClinicosDeta lle.asp?idsolicitud=1499. [Accessed Last] 25 January 2018.

- 3. Chow S, Wang H, Shao J. Sample size calculation in Clinical Research. New York: Taylor Francis, 2007.
- International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. Clinical Safety Data Management: Definitions and Standards for Expedited Reporting E2A. ICH Harmonised Tripartite Guideline, Vol. 4, 1994.
- 5. Haffajee A, Socransky S, Lindhe J. Comparison of satatistical methods of analysis of data from clinical periodontal trials. J Clin Periodontol, 1983, 247-56.
- 6. Woolson R. Wilcoxon signed-rank test. Wiley Encyclopedia of clinical trials, 2008, 1-3.

### Annexes

# Eye Comfort Index

| | E | ye Com | fort Inde | X | | |
|---|---|---|---|---|---|---|
| Identification o | | | | | | ************** |
| Study No.: SOPH1 | 72-0919-1 | | | | Date: / | 1 |
| Subject's initia | ls: | | | Subjec | t No.: 172 | |
| Directions: | | | | | | |
| | ire was designed to r | rate the comfort | of your owne | | | |
| | on, circle your answe | | oi your eyes. | | | |
| Example: | In the past week, ho | w often were yo | ur eyes red? | | | |
| | Never<br>0 1 | 2 | 3 | 4 5 | Always_<br>6 | |
| There are no rig | ht or wrong answers | . Don't spend to | o much time on | each question. | | |
| - | | | | | | |
| 1 In the p | ast week, how often | did your eyes fe | el dry ? | | | |
| Never | | | | | | Always |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 114 | | | e . | | | |
| | our eyes felt dry, how | v severe was the | e sensation usu | iany? | | Source |
| I haven't fel | 1 | 2 | 3 | 4 | 5 | Severe<br>6 |
| | | | _ | | _ | - |
| 2 In the p | ast week, how often | did your eyes fe | el gritty ? | | | |
| Never | | | | | | Alwaya |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | our eyes felt <i>gritty,</i> ty | pically, how inte | nse was the se | ensation? | | |
| I haven't fel | <u>t it</u><br>1 | 2 | 3 | 4 | 5 | Severe<br>6 |
| v | | 2 | 3 | 7 | 3 | ٥ |
| 3 In the p | ast week, how often | did vour eves fe | el throbbina ? | | | |
| Never | | , , | | | | Always |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| - | our eyes felt like <i>the</i> y | were stinging, | how intense wa | is the sensation u | isually? | |
| I haven't fel | | | | | _ | Severe |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| A In the past w | veek, how often did y | our avec feel fin | ad 2 | | | |
| Never | reak, now olleri did y | our eyes reer un | ou r | | | ****** |
| 0 | 1 | 2 | 3 | 4 | 5 | Always 6 |
| When y | When your eyes felt tired, how intense was the feeling usually? | | | | | |
| I haven't fel | | | | | | Severe |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | | | | Observed a second |

| 5 | - | eek, how often | did your eyes fee | el sore ? | | | |
|---|---|---|---|---|---|---|---|
| | <u>Never</u><br>0 | 1 | 2 | 3 | 4 | 5 | Always 6 |
| | When your e | yes felt <i>sore,</i> h | ow severe was th | e sensation us | ually? | | i |
| 1 | haven't felt it | | | | | | Severe |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 6 | In the past w | eek, how often | did your eyes fee | el itchy ? | | | 1 |
| | Never | | | | | | Always |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | When your e | yes felt <i>itchy</i> , h | now intense was t | he sensation u | sually? | | - |
| 1 | haven't felt it | | | | | | Severe |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | | | | | į |
| | | | | | | | 1 |

### Oxford Scale

| PANEL | Grade | Criteria |
|-------|-------|-----------------------------------------------|
| A | 0 | Equal to or less than panel A |
| В | I | Equal to or less than panel B, greater than A |
| С | II | Equal to or less than panel C, greater than B |
| D | III | Equal to or less than panel D, greater than C |
| E | IV | Equal to or less than panel E, greater than D |
| >E | V | Greater than panel E |